CLINICAL TRIAL: NCT03488784
Title: Natural History of Disease Progression in Individuals With Limb Girdle Muscular Dystrophy Type 2A and Type 2E
Brief Title: Natural History of Limb Girdle Muscular Dystrophy Type 2A and Type 2E
Status: Completed | Type: Observational
Sponsor: Lindsay Alfano (Other)
Responsible Party: Sponsor-Investigator, Lindsay Alfano, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB17-01086
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Limb-Girdle Muscular Dystrophy Type 2A; Limb-Girdle Muscular Dystrophy, Type 2E
MeSH Terms: conditions — Limb-girdle muscular dystrophy type 2A; Limb-girdle muscular dystrophy, type 2E

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational study, no drug (marketed or investigational) will be provided as part of the study, and the study procedures will have no impact on the medical care delivered to patients participating in this study. The overall study data collection period is planned to last up to 5 years with assessments occurring at baseline, and every 6 months thereafter for a total period of 3 years.

Medical records for enrolled patients will be abstracted at baseline and annually to obtain clinical information, and data will be recorded for the study. Eligible patients will be asked to provide informed consent and to complete semi-annual patient surveys and functional assessments. The patient surveys will include selected PRO instrument(s) along with additional questions to characterize the patient's perception of disease.

DETAILED DESCRIPTION:
Neuromuscular disease can be characterized by progressive muscle degeneration, impaired pulmonary status, and decreased cardiac function.(1-8) Additionally, these neuromuscular disorders can be rare, and therefore difficult to establish the natural progression of each disease.The natural history of each neuromuscular disorder provides valuable information about the specific progression of the disease, which can guide in understanding which outcomes to measure in order to show change for clinical trials. Experimental treatments for many of these neuromuscular disorders are currently being assessed in clinical trials with others in the pipeline for upcoming clinical trials in the near future. Thus, the need to reliably and objectively detect small, meaningful changes in daily functional activities in order to serve as a supportive measure of efficacy in clinical trials is of great importance.

Functional and strength measures have been utilized as primary, secondary or exploratory outcomes in clinical trials studying the efficacy of drug therapies. Many of these outcome measures have been shown to be reliable and have been validated in neuromuscular disease.

This longitudinal study aims to characterize the clinical progression and functional impact on patients with neuromuscular disorders over time by evaluating functional and patient-reported outcomes (PROs). The association between functional impairment and long-term outcomes, such as loss of mobility, falls, and quality of life, will be examined.

ELIGIBILITY:
Inclusion Criteria:

Suspected LGMD2A or LGMD2E by symptoms and having a family member diagnosed with 2A or 2E, or have genetic confirmation of one of these two types of LGMD themselves.

Perform assessments to the best of their ability with reliable results as deemed by the evaluator. Ability to attend scheduled appointments Ability to provide informed consent (or assent for ages 9-18)

Exclusion Criteria:

Confirmed diagnosis of neuromuscular disorder other than LGMD2E or LGMD2A Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's well being, safety, or clinical interpretability.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals suspected of having LGMD type 2E or type 2A due to symptoms and a diagnosed family member or a member of a community with a large population of one of these two types. Individuals with a diagnosis of LGMD2E or LGMD2A with genetic testing including carriers of type 2E or type 2A
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Strength | 6 months
  Force production testing using standardized equipment

SECONDARY OUTCOMES:
Walking speed | 6 months
  Timing how fast the person can walk 100 meters
Physical functioning | 6 months
  Observing or surveying how well a person can perform activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Linda Lowes, PT PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No